CLINICAL TRIAL: NCT00123669
Title: The Primary Progesterone Therapy for Operable Breast Cancer : A Randomized Controlled Trial
Brief Title: Primary Progesterone Therapy for Operable Breast Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tata Memorial Hospital (Other Government)
Collaborators: Ministry of Science and Technology, India (Other Government)
Responsible Party: Principal Investigator, Dr Rajendra A. Badwe, Director, Tata Memorial Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: No. SP/SO/B29/2000
Record Dates: First submitted 2005-07-21; First posted 2005-07-25 (Estimated); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Breast Neoplasms
Keywords: Cancer of the Breast; Neoplasm
MeSH Terms: conditions — Breast Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Patient will not receive Inj Progesterone 500 mg
- Treatment (Experimental): An intramuscular injection of 500mg depot hydroxy-progesterone 5-14 days prior to surgery.
  Interventions: Drug: 500 mg of depot hydroxy-progesterone

INTERVENTIONS:
Drug: 500 mg of depot hydroxy-progesterone — An intramuscular injection of 500 mg of depot hydroxy-progesterone 5 to 15 days prior to surgery.
  Arms: Treatment

SUMMARY:
The purpose of this study is to test the effect of primary progesterone on overall and disease free survival in women with operable breast cancer. The study addresses two issues related to breast cancer surgery:

* Circulating progesterone at the time of surgery might counteract the detrimental effect of estrogen on survival of women with operable breast cancer.
* Events at the time of surgery may have an impact on the natural history of breast cancer

DETAILED DESCRIPTION:
This protocol addresses the issue of pre-operative hormone manipulation in women with operable breast cancer. The study has been designed after careful review of literature to assess the effect of unopposed oestrogen at the time of surgery and collect evidence that events at the time of surgery may have impact on the long-term survival of breast cancer patients. The meta-analysis of 37 studies on timing of surgery during the menstrual cycle showed a 15% + 3 improvement in survival for women who had undergone surgery during the luteal phase of their menstrual cycle. Three of the 37 studies where progesterone levels were estimated at the time of surgery showed 52% + 26 improvement in survival when circulating progesterone were > 1.5 ng/ml. The study aims to produce luteal milieu by injecting Hydroxy- progesterone 500 mg IM at the time of surgery. The timing of administration of progesterone in the neo-adjuvant setting is decided after collating data from large data-bases and randomised trials of screening suggesting that events at the time of surgery may alter the behavior of micro-metastases.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral operable palpable breast cancer

Exclusion Criteria:

* Previous history of excision biopsy of the primary tumour
* History of other epithelial/mesenchymal malignant tumours except basal cell carcinoma/squamous cell carcinoma (BCC/SCC) of skin

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 1997-10; Primary Completion 2020-05-29 (Actual); Study Completion 2020-05-29 (Actual)

PRIMARY OUTCOMES:
To test the effect of primary progesterone in operable breast cancer on overall and disease free survival at 5 years | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Rajendra A Badwe, M.S., Principal Investigator — Professor & Head, Department of Surgical Oncology, Chief Breast Unit
Locations (1):
- Tata Memorial Hospital, Mumbai, Maharashtra, India

REFERENCES:
- [Background] Badwe RA, Wang DY, Gregory WM, Fentiman IS, Chaudary MA, Smith P, Richards MA, Rubens RD. Serum progesterone at the time of surgery and survival in women with premenopausal operable breast cancer. Eur J Cancer. 1994;30A(4):445-8. doi: 10.1016/0959-8049(94)90415-4. PMID 8018400
- [Background] Badwe RA, Gregory WM, Chaudary MA, Richards MA, Bentley AE, Rubens RD, Fentiman IS. Timing of surgery during menstrual cycle and survival of premenopausal women with operable breast cancer. Lancet. 1991 May 25;337(8752):1261-4. doi: 10.1016/0140-6736(91)92927-t. PMID 1674070
- [Background] Badwe RA, Bettelheim R, Millis RR, Gregory W, Richards MA, Fentiman IS. Cyclical tumour variations in premenopausal women with early breast cancer. Eur J Cancer. 1995 Dec;31A(13-14):2181-4. doi: 10.1016/0959-8049(95)00301-0. PMID 8652239
- [Background] Badwe RA, Mittra I, Havaldar R. Timing of surgery with regard to the menstrual cycle in women with primary breast cancer. Surg Clin North Am. 1999 Oct;79(5):1047-59. doi: 10.1016/s0039-6109(05)70060-8. PMID 10572550
- [Background] Badwe RA, Hawaldar RW. Effect of menstrual phase on surgical treatment of breast cancer. Lancet. 1994 Aug 6;344(8919):404. No abstract available. PMID 7914322
- [Background] Badwe RA, Juvekar RR. Timing of breast cancer surgery during the menstrual cycle. Ann Oncol. 1994 Jan;5(1):29-31. doi: 10.1093/oxfordjournals.annonc.a058682. No abstract available. PMID 8172788
- [Derived] Badwe R, Hawaldar R, Parmar V, Nadkarni M, Shet T, Desai S, Gupta S, Jalali R, Vanmali V, Dikshit R, Mittra I. Single-injection depot progesterone before surgery and survival in women with operable breast cancer: a randomized controlled trial. J Clin Oncol. 2011 Jul 20;29(21):2845-51. doi: 10.1200/JCO.2010.33.0738. Epub 2011 Jun 13. PMID 21670457